CLINICAL TRIAL: NCT07191873
Title: A Phase IV Placebo-controlled Single Center Trial for Tirzepatide in Idiopathic Intracranial Hypertension Trial (TIIHT)
Brief Title: Tirzepatide in Idiopathic Intracranial Hypertension Trial
Acronym: TIIHT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00117470
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Intracranial Hypertension (IIH)
Keywords: IIH; BMI; Eye Pressure; Headache
MeSH Terms: conditions — Pseudotumor Cerebri; Headache | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide (Active Comparator): Participants receive Tirzepatide weekly on the following dose schedule for a year:
  Dosage Treatment time 2.5mg/0.5mL: Month 1 (4 Weeks) 5mg/0.5mL: Month 2 (4 Weeks) 7.5mg/0.5mL: Month 3 (4 Weeks) 10mg/0.5mL: Month 4 (4 Weeks) 12.5mg/0.5mL: Month 5-6 15mg/0.5 mL: Month 7-12
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants receive Tirzepatide Placebo weekly on the following dose schedule for a year:
  Dosage Treatment time 2.5mg/0.5mL: Month 1 (4 Weeks) 5mg/0.5mL: Month 2 (4 Weeks) 7.5mg/0.5mL: Month 3 (4 Weeks) 10mg/0.5mL: Month 4 (4 Weeks) 12.5mg/0.5mL: Month 5-6 15mg/0.5 mL: Month 7-12
  Interventions: Drug: Tirzepatide Placebo

INTERVENTIONS:
Drug: Tirzepatide — Dosage Treatment time 2.5mg/0.5mL: 4 Weeks 5mg/0.5mL: 4 Weeks 7.5mg/0.5mL: 4 Weeks 10mg/0.5mL: 4 Weeks 12.5mg/0.5mL: 4 weeks 15mg/0.5 mL: 7 Months
  Arms: Tirzepatide
Drug: Tirzepatide Placebo — Dosage Treatment time 2.5mg/0.5mL: 4 Weeks 5mg/0.5mL: 4 Weeks 7.5mg/0.5mL: 4 Weeks 10mg/0.5mL: 4 Weeks 12.5mg/0.5mL: 4 weeks 15mg/0.5 mL: 7 Months
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, parallel, placebo-controlled trial of 60 participants. The primary analysis will be a statistical comparison of the estimates of the mean difference in the 12-month change in intracranial pressure (ICP) between participants assigned to the tirzepatide and Placebo arms in 1:1 randomization using the intention-to-treat (ITT) population. Hypothesis testing will be performed using analysis of covariance (ANCOVA), with the treatment indicator as the independent variable and the 12-month change in ICP as the dependent variable. Models will include baseline ICP as a covariate. This primary endpoint will use a significance level of 0.05 to declare significance.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms of increased intracranial pressure:

   1. headaches, tinnitus, visual obscurations, papilledema;
   2. absence of localizing findings on neurological examination (except for VI nerve palsy);
   3. no secondary causes identified on imaging, e.g., hydrocephalus, space- occupying lesion;
   4. elevated lumbar puncture (LP) opening pressure (OP) ≥25 cm H2O in lateral decubitus position with legs extended (>= (≥ 20cm H2O if one of the following is present: pulse synchronous tinnitus, abducens palsy, Frisen grade II papilledema, transverse venous sinus stenosis, partially empty sella or enlarged optic nerve sheath on magnetic resonance imaging (MRI);
   5. the patient is awake and alert.
2. BMI ≥30 kg/m2
3. Age 18-60 years of age
4. Unilateral or bilateral papilledema
5. Able to provide informed consent
6. Women of child-bearing age must use birth control (non-oral contraceptive method or add a barrier method of contraception).

Exclusion Criteria:

1. Previous bariatric surgery
2. Prior intervention for high ICP including optic nerve sheath fenestration (ONSF), venous stenting and/or shunting
3. Taking another GLP-1 agonist, another drug that can interfere with the GLP-1 agonist, or any other anti-obesity medication
4. History of pancreatitis, personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN2), history of gallbladder disease, ulcerative colitis, Crohn's disease, or history of hypersensitivity reaction in response to the drug
5. Pregnancy or planning a pregnancy in the next 12 months or currently breastfeeding
6. Other disorders causing visual loss and/or anomalous optic nerve
7. Taking another medication to lower ICP in IIH (if previously taking another medication for ICP must be off this medication for at least 30 days prior to enrollment)
8. No change in headache medications in the past 60 days
9. Venous sinus thrombosis on magnetic resonance venography (MRV)
10. Papilledema Frisen Grade III, IV or fulminant IIH
11. Mean perimetric deviation ≤ -7 dB
12. CSF contents outside of normal limits
13. Uncontrolled hypertension (≥140mmHg/90 mmHg)
14. Anemia (hemoglobin [Hgb] ≤ 8.0g/dL)
15. Diagnosed sleep apnea with continuous positive airway pressure (CPAP) use
16. Exposure to a drug, substance, or disorder that has been associated with elevation of intracranial pressure within 2 months of diagnosis such as lithium, vitamin A, various cyclines
17. eGFR < 30 ml/min/1.73m2
18. Type II diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in intracranial pressure in Idiopathic Intracranial Hypertension (IIH) patients | From enrollment to end of treatment at 12 months
  Assessed by opening pressure via lumbar puncture (LP) in the left lateral decubitus position and measured in cm H2O.

SECONDARY OUTCOMES:
Retinal Nerve Fiber Layer (RNFL) Thickness on optical coherence tomograhy (OCT) | From enrollment to end of treatment at 12 months
  Mean change in RNFL thickness
Change in Frisen papilledema grade on fundus photography | From enrollment to the end of treatment at 12 months
  The Frisen scale ranges from 0 (normal optic disc) to 5 (severe degree of edema).
Change in perimetric mean deviation | From enrollment to end of treatment at 12 months
  Perimetric Mean Deviation (MD) is a key visual field index that represents the average point-by-point difference between a patient's visual field and the normal, age-matched expected visual field.

CONTACTS AND LOCATIONS:
Overall Officials: Alexa N Bramall, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spitze A, Lam P, Al-Zubidi N, Yalamanchili S, Lee AG. Controversies: Optic nerve sheath fenestration versus shunt placement for the treatment of idiopathic intracranial hypertension. Indian J Ophthalmol. 2014 Oct;62(10):1015-21. doi: 10.4103/0301-4738.146012. PMID 25449938
- [Background] Chen J, Wall M. Epidemiology and risk factors for idiopathic intracranial hypertension. Int Ophthalmol Clin. 2014 Winter;54(1):1-11. doi: 10.1097/IIO.0b013e3182aabf11. No abstract available. PMID 24296367
- [Background] Mollan SP, Ali F, Hassan-Smith G, Botfield H, Friedman DI, Sinclair AJ. Evolving evidence in adult idiopathic intracranial hypertension: pathophysiology and management. J Neurol Neurosurg Psychiatry. 2016 Sep;87(9):982-92. doi: 10.1136/jnnp-2015-311302. Epub 2016 Feb 17. PMID 26888960
- [Background] Miah L, Strafford H, Fonferko-Shadrach B, Hollinghurst J, Sawhney IMS, Hadjikoutis S, Rees MI, Powell R, Lacey A, Pickrell WO. Incidence, Prevalence, and Health Care Outcomes in Idiopathic Intracranial Hypertension: A Population Study. Neurology. 2021 Feb 22;96(8):e1251-e1261. doi: 10.1212/WNL.0000000000011463. PMID 33472926
- [Background] Mollan SP, Aguiar M, Evison F, Frew E, Sinclair AJ. The expanding burden of idiopathic intracranial hypertension. Eye (Lond). 2019 Mar;33(3):478-485. doi: 10.1038/s41433-018-0238-5. Epub 2018 Oct 24. PMID 30356129